CLINICAL TRIAL: NCT04455399
Title: Time Efficiency Comparison of Two Intravitreal Injection Techniques
Acronym: TIVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peregrine Eye and Laser Institute (Other)
Responsible Party: Principal Investigator, Harvey Siy Uy, Medical Director, Peregrine Eye and Laser Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200102
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion With Macular Edema; Uveitic Macular Edema; Choroidal Neovascularization
Keywords: intravitreal injection; intravitreal injecton guide; macular edema; time efficiency; anti-VEGF
MeSH Terms: conditions — Choroidal Neovascularization; Macular Edema

STUDY DESIGN:
Intervention Model Description: Intravitreal Injection Guide (Malosa, Beaver Visitec International, Waltham, MA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravitreal injection guide (Other): Single use, combination ocular surface caliper to determine point of intravitreal injection and set-depth injection guide to limit injection needle entry into the eye
  Interventions: Device: Intravitreal injection guide (Malosa)
- Dual blade eyelid speculum (Other): Dual blade eyelid speculum to open eyelids followed by Castroviejo surgical caliper to measure injection point 3.5 mm from limbus
  Interventions: Device: Dual Blade Eyelid Speculum

INTERVENTIONS:
Device: Intravitreal injection guide (Malosa) — A single use, multifunction device will be used to push away an eyelid to expose injection site, indicate injection point about 4 millimeters from surgical limbus, and directs needle perpendicular to the ocular surface while limiting intraocular needle incursion
  Other Names: Malosa intravitreal injection guide
  Arms: Intravitreal injection guide
Device: Dual Blade Eyelid Speculum — A conventional dual blade eyelid speculum will be use to push away eyelids. A Castroviejo surgical caliper will be used to mark the injection site.
  Arms: Dual blade eyelid speculum

SUMMARY:
Prospective, single-center, randomized, clinical trial (RCT) comparing the time efficiency and safety of a single-use intravitreal injection (IVI) guide versus a traditional technique using a dual blade speculum among patients undergoing IVI for various indications.

DETAILED DESCRIPTION:
Prospective, single-center, randomized, clinical trial (RCT) comparing the efficiency and safety of a single-use IIG with a traditional technique using a dual blade speculum among patients undergoing IVI for various indications.

The investigators will include eyes of adult patients scheduled to undergo unilateral IVI for neovascular age-related macular degeneration (nAMD), polypoidal choroidal vasculopathy (PCV), diabetic macular edema (DME), retinal vein occlusion (RVO), choroidal neovascular membrane from pathologic myopia (PM) and uveitis. The investigators will exclude eyes with a history of extraocular or intraocular infection within 3 months of the scheduled IVI date, scleral thinning, history of previous glaucoma surgery, history of pars plana vitrectomy, hypersensitity to the IVI drug, propracaine or povidone iodine, and inability to understand the informed consent form.

The eyes will be randomly assigned in 1:1 fashion into two injection arms: intravitreal injection guide (IIG) and dual blade speculum (DBS). At the time of injection, a random number generator will be used to generate an odd or even number for each eye. Odd eyes will be assigned to IIG and even eyes will be assigned to DBS. For same day bilateral injection, once the first eye is randomized to one technique, the second eye will be automatically assigned to the other technique. The study will be conducted in compliance with the Declaration of Helsinki. All patients will provide informed consent prior to start of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Eyes of adult patients requiring intravitreally injected medications for non-infectious indications

Exclusion Criteria:

* History of extraocular or intraocular infection within 3 months of the scheduled IVI date
* Scleral thinning
* History of previous glaucoma surgery
* History of pars plana vitrectomy
* Hypersensitivity to the IVI drug, proparacaine or povidone iodine
* Inability to understand the informed consent form

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Duration of intravitreal injection procedure | At time of injection procedure
  Duration in seconds from application to removal of single-blade or dual blade speculum

SECONDARY OUTCOMES:
Adverse event rate | Immediately and up to 1 month after the intravitreal injection procedure
  Frequency of adverse events and serious adverse events after intravitreal injection
Patient preference for IVI technique | Immediately post injection using single-blade speculum
  Patient survey as to which technique is more comfortable and preferred among patients with prior injection experience using the dual blade speculum

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Uy, MD, Principal Investigator — Peregrine Eye and Laser Institute
Locations (1):
- Peregrine Eye and Laser Instittute, Makati City, MM, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uy HS, Artiaga JCM. Comparison of Two Different Intravitreal Injection Techniques. Clin Ophthalmol. 2021 Jun 8;15:2383-2389. doi: 10.2147/OPTH.S309501. eCollection 2021. PMID 34135566